CLINICAL TRIAL: NCT01060176
Title: Three Dose Regimen of Tranexamic Acid on Blood Loss and Allogeneic Transfusions in Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Three Dose Regimen of Tranexamic Acid in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Associate Professor and Vice Chair of the Department of Anesthesiology, Fuwai hospital, NCCD, PUMC & CAMS, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXA Dosage Trial
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Hemostasis
Keywords: tranexamic acid; cardiac surgery procedures; hemostasis
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High dosage (Experimental): Tranexamic acid with a loading dose of 30 mg/kg and a maintenance infusion of 20 mg/kg/h
  Interventions: Drug: Tranexamic Acid
- Medium dosage (Experimental): Tranexamic acid with a loading dose of 20 mg/kg and a maintenance infusion of 15 mg/kg/h
  Interventions: Drug: Tranexamic Acid
- Low dosage (Experimental): Tranexamic acid with a loading dose of 10 mg/kg and a maintenance infusion of 10 mg/kg/h
  Interventions: Drug: Tranexamic Acid
- Control (Placebo Comparator): Saline solution
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: High dosage; Low dosage; Medium dosage
Drug: Saline Solution
  Arms: Control

SUMMARY:
Tranexamic acid is thought to be a promising substitute for aprotinin when the latter has seceded in 2007. Yet the ideal dosage and dosing regimen of tranexamic acid in cardiopulmonary bypass cardiac surgery in Chinese population remains controversial. The current study includes patients receiving valvular replacement and coronary artery bypass surgery. Three dosage regimen of tranexamic acid is delivered and blood loss, transfusions and clinical outcomes are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatic or recessive valvular disease patients requiring valvular replacement surgery with cardiopulmonary bypass
* Coronary artery disease patients requiring coronary artery bypass surgery with cardiopulmonary bypass
* Wrriten consent obtained

Exclusion Criteria:

* Non-primary cardiac surgery
* Preoperative liver or renal dysfunction
* Preoperative coagulation disorder
* Allergy
* Pregnancy or lactation
* Disabled in spirit or law
* Fatal conditions such as tumour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of exposure to allogeneic erythrocytes transfusions | Perioperatively
  Allogeneic RBCs were transfused if the hemoglobin level was less than 6 g/dL during cardiopulmonary bypass, less than 8 g/dL postoperatively, or less than 9 g/dL for elderly people (>70 years).

SECONDARY OUTCOMES:
Volume of allogeneic erythrocytes transfusions | Perioperatively
  Allogeneic RBCs were transfused if the hemoglobin level was less than 6 g/dL during cardiopulmonary bypass, less than 8 g/dL postoperatively, or less than 9 g/dL for elderly people (>70 years).
Rate and volume of fresh frozen plasma transfusion | Perioperatively
Rate and volume of allogeneic platelet transfusion | Perioperatively
Rate of reexploration for hemostasis | Perioperatively
Postoperative blood loss | Postoperatively
  Defined as total volume of chest drainage postoperatively
Thromboelastography | Perioperatively
Coagulatory and fibrinolytic associated moleculars | Perioperatively
  FIB, FDP, FXI:C, AT-III, D-dimer and TXB2
Inflammation associated moleculars | Perioperatively
  ET-1, IL-2, IL-6, IL-8, IL-10, TNF-α, NE, FN and PGI2
Length of stay in ICU and hospital postoperatively | Postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Lihuan Li, MD, Study Chair — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC; Jia Shi, MD, Principal Investigator — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China